CLINICAL TRIAL: NCT05796739
Title: SMart Angioplasty Research Team-Pragmatic Randomized Trial for Comparing Routine Versus As-Needed EXercise or Pharmacologic Stress Testing in Asymptomatic Patients With High-Risk Coronary CalciuM (SMART-EXAM)
Brief Title: Routine Versus As-Needed Stress Testing in Asymptomatic Patients With High-Risk Coronary Calcium
Acronym: SMART-EXAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung-Hyuk Choi, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SMART-EXAM
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Coronary Atherosclerosis Due to Calcified Coronary Lesion
Keywords: Non-invasive stress test; Coronary calcification; Agatston score

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine stress testing (Experimental): In this group, the preselected functional stress testing (exercise electrocardiography, stress echocardiography, nuclear imaging, or stress cardiac magnetic resonance imaging) will be performed within three months (± 2 months) according to the practice pattern of each participating center.
  Interventions: Diagnostic Test: Non-invasive stress test
- As-needed stress testing (Active Comparator): In this group, optimal medical treatment will be performed by current guidelines without further testing. A stress test will be performed only when new symptoms (exertional chest pain or dyspnea) occur that may clinically suggest significant coronary artery disease.
  Interventions: Diagnostic Test: Medical treatment without further testing

INTERVENTIONS:
Diagnostic Test: Non-invasive stress test — Nuclear imaging, stress echocardiography, exercise electrocardiography, stress cardiac magnetic resonance imaging
  Arms: Routine stress testing
Diagnostic Test: Medical treatment without further testing — Optimal medical treatment for primary prevention.
  Arms: As-needed stress testing

SUMMARY:
The purpose of the SMART-EXAM (SMart Angioplasty Research Team-Pragmatic Randomized Trial for Comparing Routine versus As-Needed EXercise or Pharmacologic Stress Testing in Asymptomatic Patients with High-Risk Coronary CalciuM) trial is to compare the major adverse cardiovascular events between routine stress testing and as-needed stress testing in asymptomatic patients with high-risk coronary calcium (Agatston Score ≥ 400) without proven ASCVD.

DETAILED DESCRIPTION:
The coronary artery calcium (CAC) scan, a marker of subclinical coronary atherosclerosis, has become popular for individuals at risk for atherosclerotic cardiovascular disease. CAC is strongly associated with atherosclerotic burden and predicts coronary heart disease events and mortality, regardless of their age, sex, race, or atherosclerotic cardiovascular disease (ASCVD) risk. Furthermore, the progression of CAC is associated with an increased risk for future hard and total coronary heart disease events. The use of CAC scoring was associated with significant improvements in the reclassification and discrimination of incident ASCVD. Nevertheless, the current guidelines recommend CAC measurement for selected cases only with borderline or intermediate risk of ASCVD. However, in real-world practice, CAC testing is increasingly being promoted to the public as a means of self-assessment of cardiovascular risk and is widely being used regardless of ASCVD risk.

Non-invasive stress testing is often recommended to exclude potentially dangerous coronary artery disease. However, stress testing in asymptomatic individuals has low sensitivity and specificity.9 Although the 2019 Primary Prevention of Cardiovascular Disease Guidelines do not comment on functional or invasive testing in asymptomatic individuals with a high CAC score, the 2009 Appropriate Use Criteria for Cardiac Radionuclide Imaging report gives a level A recommendation for obtaining a stress test in asymptomatic individuals with CAC score ≥400.10 In addition, the 2013 update of the 2009 document also considers stress imaging appropriate for patients with CAC score >100. However, there have been no large randomized controlled trials or observational studies that have evaluated the utility of functional or invasive testing in asymptomatic individuals free of ASCVD with high CAC scores. Theoretically, early detection and revascularization of ischemia producing lesions in asymptomatic patients with high-risk coronary calcification without proven ASCVD might reduce the future risk of major adverse cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 19 years of age. ② Asymptomatic patients with high-risk coronary calcium (Agatston Score ≥ 400)

Exclusion Criteria:

* Documentation of objective evidence of inducible ischemia before enrollment

  * Presence of significant coronary artery stenosis (≥ 70% diameter stenosis) confirmed by coronary angiography or coronary computed tomography angiography before enrollment

    * History of coronary revascularization procedure ④ Pregnancy or breast feeding ⑤ Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment) ⑥ Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of major adverse cardiovascular events | up to 4.5 years of median follow-up
  a composite of death from cardiovascular causes, myocardial infarction, unplanned hospitalization leading to an urgent revascularization procedure, or heart failure hospitalization

SECONDARY OUTCOMES:
cardiovascular death | up to 4.5 years of median follow-up
  death from cardiovascular causes
myocardial infarction | up to 4.5 years of median follow-up
  myocardial infarction
unplanned hospitalization leading to an urgent revascularization procedure | up to 4.5 years of median follow-up
  unplanned hospitalization leading to an urgent revascularization procedure
heart failure hospitalization | up to 4.5 years of median follow-up
  heart failure hospitalization
all-cause death | up to 4.5 years of median follow-up
  death from any causes
a composite of death from cardiovascular cause or myocardial infarction | up to 4.5 years of median follow-up
  a composite of death from cardiovascular cause or myocardial infarction
any hospitalization | up to 4.5 years of median follow-up
  any hospitalization
performing revascularization procedure | up to 4.5 years of median follow-up
  performing revascularization procedure
performing invasive coronary angiography procedure | up to 4.5 years of median follow-up
  performing invasive coronary angiography procedure
stroke | up to 4.5 years of median follow-up
  stroke
bleeding | up to 4.5 years of median follow-up
  Bleeding Academic Research Consortium type 2-5
total medical cost | up to 4.5 years of median follow-up
  total medical cost

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hyuk Choi, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- SamsungMedicalCenter, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided